CLINICAL TRIAL: NCT02507778
Title: Circulating Tumor Cells Spillage After Pulmonary Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Nir Peled, Professor, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0468-14-RMC
Record Dates: First submitted 2015-07-14; First posted 2015-07-24 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: Lung; Cancer; Biomarkers; Early detection; Circulating tumor cell
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Neoplastic Cells, Circulating | interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biopsy (Other): needle will be inserted before and after biopsy and will measure circulating tumor cells.
  Interventions: Device: CellCollectorTM (Gilupi, Germany) needle

INTERVENTIONS:
Device: CellCollectorTM (Gilupi, Germany) needle — needle will be inserted before and after biopsy and will measure circulating tumor cells.

SUMMARY:
The aim of this study is to quantify the spillage of tumor cells after biopsy in early lung cancer.

DETAILED DESCRIPTION:
Introduction:

Lung cancer (NSCLC) is a common malignancy with a high recurrence rate even when diagnosed at early stages. Biopsy is currently the procedure of choice for the investigation of pulmonary lesions, yet it is unclear whether the biopsy itself releases tumor cells into the circulation and attributes to the late distal recurrence.

Studies of various malignancies show the ability to identify circulating tumor cells (CTCs) even in early stage cancer. The number of CTCs correlates with disease outcome. Dynamics of CTCs after CT or bronchoscopy guided biopsy has not been evaluated so far. In the metastatic setting, the number of CTCs correlates to tumor response to chemotherapy in both small and non-small lung cancer (SCLC and NSCLC, respectively).

The aim of this study is to quantify the spillage of tumor cells after biopsy in early lung cancer.

Patients with suspected pulmonary lesions undergoing CT or bronchoscopy guided biopsy will be enrolled into the study. The CellCollectorTM will be used for CTCs detection before and after the procedure. These patients will be their own controls.

In this study the investigators will use the CellCollectorTM (Gilupi, Germany) needle that isolates CTCs of epithelial origin using a needle coated with antibodies directed against the epithelial cell adhesion molecules (EpCAM). This technology enables high quality immunohistochemical and molecular testing of the acquired cells as needed for treatment planning, and even allows cell culture growth from the live CTCs. This device is certified for use throughout Europe, with no adverse events noted with its usage .

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of lung cancer
* Patients are designated to undertake biopsy
* Able and willing to participate in this study
* Availability of a signed informed consent

Exclusion Criteria:

* Any recent non-lung cancer in the recent 2 years.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor cells (CTCs) before and after the procedure. | 1 day
  In this study we will use for CTC counting the CellCollectorTM (Gilupi, Germany) needle that isolates CTCs of epithelial origin using a needle coated with antibodies directed against the epithelial cell adhesion molecules (EpCAM).

CONTACTS AND LOCATIONS:
Overall Officials: Nir Peled, MD PhD FCCP, Principal Investigator — nirp@clalit.org.il
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No